CLINICAL TRIAL: NCT03324854
Title: Use of Mosquito Net Mesh in Comparison With Polypropylene Mesh for Ventral Hernia Repair.
Brief Title: Use of Mosquito Net Mesh for Ventral Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, David Esmer, Head of general surgery, Department of surgery, Hospital Central "Dr. Ignacio Morones Prieto"
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1721
Record Dates: First submitted 2017-10-18; First posted 2017-10-30 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Hernia, Ventral; Ventral Incisional Hernia
Keywords: Mosquito net; Mesh; Polypropylene mesh; Prolene mesh; ventral hernia; hernia
MeSH Terms: conditions — Hernia, Ventral; Hernia | interventions — Drainage

STUDY DESIGN:
Intervention Model Description: The simple size for pilot study was been calculated in 20 patients, according with Browne for not knowing the variability of the treatment. 10 patients in the group of Polypropylene mesh (Prolene ®) and , and 10 patients in the group of mesh of PEBD (mosquito net).
Who Masked: Participant, Outcomes Assessor
Masking Description: The randomisation for allocation the type of mesh for each patient was realized with numbers generated by computer with the program R version 3.0.2 with the simple function.
  The participant and the outcomes assessor did not know the type of mesh.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mosquito net mesh (Experimental): The open ventral hernia repair were carried out with rives technique, followed by the placement of the mosquito net mesh, and left active-close drainage, 30 minutes before the incisión, prophylactic antibiotic 1gm of cefalotin was administered.
  Interventions: Procedure: Rives technique; Procedure: Drainage; Drug: Prophylactic
- prolene mesh (Active Comparator): The open ventral hernia repair were carried out with rives technique, followed by the placement of the prolene mesh, and left active-close drainage, 30 minutes before the incisión, prophylactic antibiotic 1gm of cefalotin was administered.
  Interventions: Procedure: Rives technique; Procedure: Drainage; Drug: Prophylactic

INTERVENTIONS:
Procedure: Rives technique — Open ventral hernia repair followed by the placement of the mesh.
Procedure: Drainage — Placement of active-close drainage in surgical site.
Drug: Prophylactic — Prophylactic antibiotic 1gm of cefalotin was administered 30 minutes before the incisión.
  Other Names: Prevention

SUMMARY:
It´s a pilot study, randomized, realized in the Central Hospital "Dr. Ignacio Morones Prieto", SLP, Mexico.

Hypothesis:

The polyethylene mesh is secure in open ventral repair.

DETAILED DESCRIPTION:
It´s a pilot study, randomized, realized in the Central Hospital "Dr. Ignacio Morones Prieto", SLP, Mexico.

The simple size for pilot study was been calculated in 20 patients, according with Browne for not knowing the variability of the treatment. 10 patients in the group of Polypropylene mesh (Prolene ®), braided monofilament thread, macropore, weight of 108.1 g/m2, fibres diameter of 0.53 mm, tensile force of 156.6 N/cm, with a pore of 1.6 mm2, in different size of 15 x 15 cm, 20 x 20 cm and 30 x 30 cm, and 10 patients in the group of mesh of PEBD (mosquito net), braided monofilament thread, macropore, ,weight of 53.7 g/m2, fibers diameter of 0.48 mm, tensile force of 42.7 N/cm and pore of 1.8 mm2, in different size 15 x 15 cm, 20 x 20 cm and 30x 30 cm donated by Dr. Ravindranath R. Tongaonkar. The sterilization were done in ethylene oxide.

The randomisation for allocation the type of mesh for each patient was realized with numbers generated by computer with the program R version 3.0.2 with the simple function.

The statistical analysis was carried out by the programs: JMP 8 (SAS Institute Inc., Cary, NC, USA) and R 2.15.1 23.

The ventral hernia repair were carried out with standardized technique, placed the mesh int the preperitoneal or retromuscular space fixing with 2-0 poplypropylene suture and le fe active-close drainage, 30 minutes before the incision, prophylactic antibiotic 1gm of cefalotin was administered, in both groups, the patient was discharge at the first postoperatory day with drainage and retired at the first review at 1 week and recited at one, three, six and twelve months for reviewer.

The descriptive analysis of categorical variables was expressed with frequencies and percentages; the numerical ones with normal distribution in averages and standard deviation, the variables with distribution not normal with medians and status (maximum and minimal values). The values of p<0.05 were considered to be significant.

This study was evaluated and accepted by the Committee of Investigation and the Committee of Ethics, with number of record 42-17.

ELIGIBILITY:
Inclusion Criteria:

* All the patients with primary or incisional elective ventral hernia repair with mesh were included, with ASA I,II and III between 18 and 75 years, of any sex, and that they accepted to take part in the protocol and signed the informed assent.

Exclusion Criteria:

* We excluded patients with incarcerated, strangulated hernia, signs of intestinal obstruction, consumption of anticoagulants, IMC >35, parastomal hernias, hernia repair with intestinal reconnections at the same procedure or presented infection in abdominal wall.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Recurrence | One year
  Rate of Reappearance of a ventral hernia post procedure after a year.

SECONDARY OUTCOMES:
Infection | first week, 1 month, 3 month, 6 month and One year
  Number of participants with open ventral hernia repair that have adverse events as infection post procedure determined by clinical, leukocytosis and positive bacterial culture.
Seroma | first week, 1 month, 3 month, 6 month and One year
  A seroma is a collection of fluid that builds up under the surface of your skin.
length of hospital stay | Days
  the average number of days that patients spend in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus M Sanchez, MD, Study Director — Universidad autonoma de san luis potosi

IPD SHARING:
Plan to Share IPD: No
As a preliminary study, its not finish yet.

REFERENCES:
- [Result] Sorensen CG, Rosenberg J. The use of sterilized mosquito nets for hernioplasty: a systematic review. Hernia. 2012 Dec;16(6):621-5. doi: 10.1007/s10029-012-0973-7. Epub 2012 Aug 3. PMID 22864684
- [Result] Tangaokar RR, Sanders DL, Kingsnorth AN (2013) Ten-Year Personal Experience of Using Low Density Polyethylene (LDPE) Mesh for Inguinal Hernia Repair. Trop Med Surg 1: 136. doi:10.4172/2329-9088.1000136
- [Result] Lofgren J, Nordin P, Ibingira C, Matovu A, Galiwango E, Wladis A. A Randomized Trial of Low-Cost Mesh in Groin Hernia Repair. N Engl J Med. 2016 Jan 14;374(2):146-53. doi: 10.1056/NEJMoa1505126. PMID 26760085
- [Result] Gundre NP, Iyer SP, Subramaniyan P. Prospective randomized controlled study using polyethylene mesh for inguinal hernia meshplasty as a safe and cost-effective alternative to polypropylene mesh. Updates Surg. 2012 Mar;64(1):37-42. doi: 10.1007/s13304-011-0103-6. Epub 2011 Aug 18. PMID 21850553
- [Result] Stephenson BM, Kingsnorth AN. Safety and sterilization of mosquito net mesh for humanitarian inguinal hernioplasty. World J Surg. 2011 Sep;35(9):1957-60. doi: 10.1007/s00268-011-1176-6. PMID 21713575
- [Result] Tongaonkar RR, Reddy BV, Mehta VK et al (2003) Preliminary multicentric trial of cheap indigenous mosquito-net cloth for tension free hernia repair. Indian J Surg 65:89-95
- [Result] Stephenson BM, Kingsnorth AN. Inguinal hernioplasty using mosquito net mesh in low income countries: an alternative and cost effective prosthesis. BMJ. 2011 Dec 15;343:d7448. doi: 10.1136/bmj.d7448. No abstract available. PMID 22174320
- [Result] Sanders DL, Kingsnorth AN, Stephenson BM. Mosquito net mesh for abdominal wall hernioplasty: a comparison of material characteristics with commercial prosthetics. World J Surg. 2013 Apr;37(4):737-45. doi: 10.1007/s00268-012-1900-x. PMID 23340707
- [Result] Sanders DL, Kingsnorth AN, Moate R, Steer JA. An in vitro study assessing the infection risk of low-cost polyethylene mosquito net compared with commercial hernia prosthetics. J Surg Res. 2013 Aug;183(2):e31-7. doi: 10.1016/j.jss.2013.01.047. Epub 2013 Feb 15. PMID 23485076
- [Result] Sanders DL, Kingsnorth AN. Operation hernia: humanitarian hernia repairs in Ghana. Hernia. 2007 Oct;11(5):389-91. doi: 10.1007/s10029-007-0238-z. Epub 2007 Jun 12. PMID 17562124
- [Result] Wilhelm TJ, Freudenberg S, Jonas E, Grobholz R, Post S, Kyamanywa P. Sterilized mosquito net versus commercial mesh for hernia repair. an experimental study in goats in Mbarara/Uganda. Eur Surg Res. 2007;39(5):312-7. doi: 10.1159/000104402. Epub 2007 Jun 25. PMID 17595545
- [Result] Wiessner R, Kleber T, Ekwelle N, Ludwig K, Richter DU. In-vitro examination of the biocompatibility of fibroblast cell lines on alloplastic meshes and sterilized polyester mosquito mesh. Hernia. 2017 Jun;21(3):407-416. doi: 10.1007/s10029-016-1550-2. Epub 2016 Nov 23. PMID 27878640
- [Result] Sharma M, Sharma DB, Chandrakar SK, Sharma D. Histopathological Comparison of Mosquito Net with Polypropylene Mesh for Hernia Repair: An Experimental Study in Rats. Indian J Surg. 2015 Dec;77(Suppl 2):511-4. doi: 10.1007/s12262-013-0904-6. Epub 2013 Apr 25. PMID 26730055
- [Result] Ambroziak A, Szepietowska K, Lubowiecka I. Mechanical properties of mosquito nets in the context of hernia repair. Comput Methods Biomech Biomed Engin. 2016 Feb;19(3):286-296. doi: 10.1080/10255842.2015.1016004. Epub 2015 Mar 10. PMID 25756655
- [Result] Patterson T, Currie P, Patterson S, Patterson P, Meek C, McMaster R. A systematic review and meta-analysis of the post-operative adverse effects associated with mosquito net mesh in comparison to commercial hernia mesh for inguinal hernia repair in low income countries. Hernia. 2017 Jun;21(3):397-405. doi: 10.1007/s10029-017-1608-9. Epub 2017 Apr 13. PMID 28409276
- [Result] Koziel S, Mitura K, Papaj P, Lorenc Z. Tension-Free Mosquito Net Mesh Inguinal Hernioplasty - an Alternative Exclusively for the Third World? Pol Przegl Chir. 2015 Feb;87(2):102-7. doi: 10.1515/pjs-2015-0027. No abstract available. PMID 26146103